CLINICAL TRIAL: NCT01983241
Title: A Randomized, Double-Blind, Placebo Controlled Study to Assess the Efficacy and Safety of Two Dose Regimens (60 mg/kg and 120 mg/kg) of Weekly Intravenous Alpha1 Proteinase Inhibitor (Human) in Subjects With Pulmonary Emphysema Due to Alpha1 Antitrypsin Deficiency
Brief Title: Efficacy and Safety of Alpha1-Proteinase Inhibitor (Human), Modified Process (Alpha-1 MP) in Subjects With Pulmonary Emphysema Due to Alpha1 Antitrypsin Deficiency (AATD)
Acronym: SPARTA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GTi1201
Record Dates: First submitted 2013-10-28; First posted 2013-11-13 (Estimated); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Emphysema in Alpha-1 PI Deficiency
Keywords: Pulmonary Emphysema; Alpha-1 Antitrypsin Deficiency; AATD; Alpha-1 PI Deficiency; Alpha-1 Proteinase Inhibitor
MeSH Terms: conditions — Pulmonary Emphysema; alpha 1-Antitrypsin Deficiency | interventions — Mp alpha1 receptor; Sodium Chloride; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alpha-1 MP 60 mg/kg (Experimental): Alpha-1 MP 60 mg/kg administered weekly by IV infusion for 156 weeks
  Interventions: Biological: Alpha-1 MP
- Alpha-1 MP 120 mg/kg (Experimental): Alpha-1 MP 120 mg/kg administered weekly by IV infusion for 156 weeks
  Interventions: Biological: Alpha-1 MP
- Placebo (Placebo Comparator): 0.9% Sodium Chloride for Injection, USP, administered weekly by IV infusion for 156 weeks
  Interventions: Other: 0.9% Sodium Chloride for Injection, USP

INTERVENTIONS:
Biological: Alpha-1 MP
  Other Names: Prolastin-C
  Arms: Alpha-1 MP 120 mg/kg; Alpha-1 MP 60 mg/kg
Other: 0.9% Sodium Chloride for Injection, USP
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, placebo-controlled, double blind clinical study to assess the efficacy and safety of two separate dose regimens of Alpha-1 MP versus placebo for 156 weeks (i.e., 3 years) using computed tomography (CT) of the lungs as the main measure of efficacy. The two Alpha-1 MP doses to be tested are 60 mg/kg and 120 mg/kg administered weekly by IV infusion for 156 weeks. The study consists of an optional pre-screening phase, Screening Phase, a 156-week Treatment Phase, and an End of Study Visit at Week 160.

ELIGIBILITY:
Inclusion Criteria:

* Have a documented total alpha1-PI serum level < 11 µM.
* Have a diagnosis of congenital AATD with an allelic combination of ZZ, SZ, Z(null), (null)(null), S(null), or "at-risk" alleles.
* At the Screening (Week -3) Visit, have a post-bronchodilator forced expiratory volume in 1 second (FEV1) ≥ 30% and < 80% of predicted and FEV1/forced vital capacity (FVC) < 70% (Global Initiative for Chronic Obstructive Lung Disease [GOLD] stage II or III).
* Have a carbon monoxide diffusing capacity (DLCO) ≤ 60% of predicted (corrected for HgB) within the past 2 years OR evidence of pulmonary emphysema on CT scan within the past 2 years per the Investigator's judgment.
* Have clinical evidence of pulmonary emphysema per the Investigator's judgment.

Exclusion Criteria:

* Has received alpha1-PI augmentation therapy for more than 1 month within the six months prior to the Screening Visit.
* Has received alpha1-PI augmentation therapy within one month of the Screening Visit.
* Has had a chronic obstructive pulmonary disease (COPD) exacerbation within the 5 weeks prior to the Screening Visit or during the Screening Phase.
* Unable to physically (e.g., unable to fit inside the CT scanner) or mentally (e.g., claustrophobic) undergo a CT scan.
* History of lung or liver transplant.
* Any lung surgery during the past 2 years (excluding lung biopsy).
* On the waiting list for lung surgery, including lung transplant.
* Smoking during the past 12 months or a positive urine cotinine test at screening that is due to smoking. Maybe on Nicotine replacement, including vapor cigarettes.
* History of anaphylaxis or severe systemic response to any plasma-derived alpha1-PI preparation or other blood product(s).
* Use of systemic steroids above a stable dose equivalent to 5 mg/day prednisone (i.e., 10 mg every 2 days) within the 5 weeks prior to the Screening Visit (inhaled steroids are not considered systemic steroids) or during the Screening Phase.
* Use of systemic or aerosolized antibiotics for a COPD exacerbation within the 5 weeks prior to the Screening Visit or during the Screening Phase.
* Known selective or severe Immunoglobulin A (IgA) deficiency.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Whole lung PD15 (15th percentile point) | Week -3 (baseline measure), Week 52, Week 104, Week 130, Week 156
  Whole lung PD15 measured by CT scan

SECONDARY OUTCOMES:
Adverse Events (AEs) | Week -3 through Week 160
  Monitoring of AEs
Serious Adverse Events (SAEs) | Week -3 through Week 160
  Monitoring of SAEs
Discontinuations from the study due to AEs | Week -3 through Week 160
  Monitoring of discontinuations due to AEs
Severe COPD Exacerbations | Week -3 through Week 160
  Severe COPD exacerbations as defined by American Thoracic Society/European Respiratory Society (ATS/ERS) criteria (i.e., COPD exacerbations requiring hospitalization)
Change from Baseline in PD15 of the basal lung region | Week -3 (baseline measure), Week 52, Week 104, Week 130, Week 156
  PD15 of the basal lung region measure by CT scan
Change from baseline in carbon monoxide diffusing capacity (DLco) | Weeks 26, 52, 78, 104, 130 and 156
  DLco performed according to American Thoracic Society/European Respiratory Society (ATS/ERS) guidelines
Changes from baseline in forced expiratory volume in 1 second (FEV1) | Weeks 26, 52, 78, 104, 130 and 156
  FEV1 performed according to ATS/ERS guidelines
Change from baseline in Saint George's Respiratory Questionnaire: Minimum value = 0, maximum value = 100, higher scores indicate worse condition | Weeks 26, 52, 78, 104, 130 and 156
  Health-related quality of life assessment tool
Change from baseline in the EuroQoL (Quality of Life)- 5 Dimension- 5 Level (EQ-5D-5L): Minimum value (for each one of the 5 levels) = 1, maximum value (for each one of the 5 levels) = 5, higher scores indicate worse condition | Weeks 26, 52, 78, 104, 130 and 156
  Heath-related quality of life assessment tool

CONTACTS AND LOCATIONS:
Locations (52):
- United States (10):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University of Florida, Gainesville, Florida
  - Medical Research of Central Florida, LLC, Leesburg, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - Accellacare, Wilmington, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Penn State Univ. Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Health Center at Tyler, Tyler, Texas
- Argentina (2):
  - Hospital del Torax Dr. Antonio A. Cetrangolo, Vicente López, Buenos Aires
  - Centro Dr. Lazaro Langer, Córdoba
- Australia (5):
  - St Vincent's Hospital Sydney, Sydney, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Institute for Respiratory Health Inc, Nedlands, Western Australia
- Brazil (3):
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - UNIFESP - Universidade Federal de São Paulo, São Paulo, São Paulo
  - Instituto do Coração - Incor- HCFMUSP, São Paulo
- Canada (3):
  - Health Sciences Centre, St. John's, Newfoundland and Labrador
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Inspiration Research Limited, Toronto, Ontario
- Denmark (2):
  - Århus Universitetshospital, Arhus C
  - Gentofte Hospital, Hellerup
- Estonia (2):
  - North Estonia Medical Centre Foundation, Tallinn
  - Tartu University Hospital, Tartu
- Turku University Central Hospital, Department of Pulmonary Diseases, Turku, Finland
- France (2):
  - Groupe Hospitalier Sud - Hôpital Haut-Lévêque, Pessac, Gironde
  - Hôpital Cardio-Vasculaire et Pneumologique Louis Pradel, Bron, Rhone
- Germany (4):
  - Universitaetsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Giessen und Marburg GmbH, Marburg, Hesse
  - Ruhrlandklinik, Essen, North Rhine-Westphalia
  - Univer des Saarlandes Innere, Homburg Saar
- Institutul de Ftiziopneumologie "Chiril Draganiuc", Chisinau, Moldova
- New Zealand (3):
  - New Zealand Respiratory and Sleep institute, Auckland
  - Christchurch Hospital NZ, Christchurch
  - Waikato Hospital, Hamilton
- Poland (2):
  - SPZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - Instytut Gruzlicy i Chorob Pluc w Warszawie, Warsaw
- Romania (2):
  - Clinic Dr.G Curteanu Oradea, Oradea
  - Spitalul Clinic de Boli Infectioase si Pneumoftiziologie, Timișoara
- Russia (3):
  - SBEI HPE Altai State Medical University of MoH and SD, Barnaul
  - FSI Scientific Research Institute of Pulmonology, Moscow
  - SAIH of Yaroslavl region "Clinical Hospital of Emergency Medical Care n.a. N. V. Solovyev, Yaroslavl
- Spain (2):
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital de Cruces, Barakaldo, Vizcaya
- Sweden (5):
  - Sahlgrenska Sjukhuset, Gothenburg
  - CTC - Clinical Trial Consultants AB, Linköping
  - Skånes Universitetssjukhus, Malmö, Malmo
  - Karolinska Universitetssjukhuset, Solna, Stockholm
  - CTC Clinical Trial Consultants AB, Uppsala

REFERENCES:
- [Derived] Sorrells S, Camprubi S, Griffin R, Chen J, Ayguasanosa J. SPARTA clinical trial design: exploring the efficacy and safety of two dose regimens of alpha1-proteinase inhibitor augmentation therapy in alpha1-antitrypsin deficiency. Respir Med. 2015 Apr;109(4):490-9. doi: 10.1016/j.rmed.2015.01.022. Epub 2015 Feb 13. PMID 25727857